CLINICAL TRIAL: NCT06405425
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of BL-B01D1 + PD-1 Combination Therapy in Patients With Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: A Study of BL-B01D1 + PD-1 in Patients With Locally Advanced or Metastatic Urothelial Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-204-03
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-B01D1 + PD-1 (Experimental): Participants receive BL-B01D1 + PD-1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1; Drug: PD-1

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: PD-1 — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This study is a phase II clinical study to explore the efficacy and safety of BL-B01D1 + PD-1 combination therapy in patients with locally advanced or metastatic urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects voluntarily participated in the study and signed informed consent;
2. Male or female aged ≥18 years and ≤75 years;
3. Expected survival time ≥3 months;
4. ECOG 0-1;
5. Unresectable locally advanced or metastatic urothelial carcinoma confirmed by histopathology and/or cytology;
6. Participants should not have received previous systemic therapy for locally advanced or metastatic urothelial cancer;
7. A biopsy sample of archived tumor tissue or metastatic urothelial carcinoma must be available within 3 years for PD-L1 and other testing;
8. At least one measurable lesion meeting the RECIST v1.1 definition was required;
9. The level of organ function must meet the requirements on the premise that blood transfusion and the use of any cell growth factors and/or platelet-raising drugs are not allowed within 14 days before the first dose;
10. Previous treatment-related toxicity returned to ≤ grade 1 defined by NCI-CTCAE v5.0;
11. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before the initiation of treatment, the serum or urine pregnancy test must be negative, and the patient must not be lactating; All enrolled patients should take adequate barrier contraception during the entire treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Prior ADC recipients with TOPI inhibitors as toxin;
2. Palliative radiotherapy within 2 weeks before the first dose;
3. Prior immunotherapy with grade ≥3 irAE or grade ≥2 immune-related myocarditis;
4. Use of an immunomodulatory drug within 14 days before the first dose of study drug;
5. The history of severe cardiovascular and cerebrovascular diseases in the past six months was screened;
6. QT prolongation, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
7. Active autoimmune and inflammatory diseases;
8. Receiving &gt before the first dose; Long-term systemic corticosteroid therapy with prednisone 10mg/d;
9. Other malignant tumors that progressed or required treatment within 5 years before the first dose;
10. Presence of: a) poorly controlled diabetes mellitus before starting study treatment; b) severe complications associated with diabetes mellitus; c) a glycated hemoglobin level of 8% or more; d) hypertension poorly controlled by two antihypertensive drugs; e) history of hypertensive crisis or hypertensive encephalopathy;
11. History of ILD, current ILD, or suspected ILD;
12. Complicated with pulmonary diseases leading to clinically severe respiratory impairment;
13. Screening for unstable thrombotic events requiring therapeutic intervention within the preceding 6 months; Infusion-related thrombosis was excluded;
14. Patients with active central nervous system metastases;
15. Patients with massive or symptomatic effusions or poorly controlled effusions;
16. Patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or allergic to any excipients of the test drug;
17. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
18. HIV antibody positive, active tuberculosis, active hepatitis B virus infection, or active hepatitis C virus infection;
19. Serious infection within 4 weeks before the first dose of study drug; Signs of pulmonary infection or active pulmonary inflammation within 4 weeks;
20. Participated in another clinical trial within 4 weeks before the first dose;
21. Patients with superior vena cava syndrome should not be rehydrated;
22. Have a history of psychotropic substance abuse with an inability to quit or a history of severe neurological or psychiatric illness;
23. Imaging examination showed that the tumor had invaded or wrapped the large thoracic vessels;
24. Severe unhealed wound, ulcer, or fracture within 4 weeks before signing the informed consent;
25. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
26. Subjects who are scheduled to receive live vaccine or receive live vaccine within 28 days before the first dose;
27. Other circumstances considered by the investigator to be inappropriate for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-B01D1 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of BL-B01D1 will be investigated.
Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-B01D1 prior to the next dose will be administered.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China